CLINICAL TRIAL: NCT07202169
Title: Pattern of the Intramural Spread of Ultralow Rectal Cancer With the Resection Margin.
Brief Title: Study of Intramural Spread Pattern in Low Rectal Cancer.
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: KY2025-R091
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Rectal Cancer Patients; Rectal Cancer Stage

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patients with T1 ultra-low rectal cancer
- Patients with T2 ultra-low rectal cancer
- Patients with T3 ultra-low rectal cancer
- Patients with T4 ultra-low rectal cancer

SUMMARY:
The purpose of this study is to study the law of intramural diffusion of low rectal cancer in different stages, and to explore the relationship between intramural diffusion of low rectal cancer and the distal resection margin during operation, so as to provide theoretical basis for clinicians to formulate accurate and individualized treatment plans, and help improve the prognosis and quality of life of patients.

ELIGIBILITY:
* Inclusion criteria

  1. Patients aged 18-75 years old
  2. Pathology suggestive of moderately to highly differentiated rectal adenocarcinoma
  3. Tumor lower margin ≤ 5 cm from the anal verge
  4. No distant metastasis such as lung, liver and other organs
* exclusion criteria

  1. Preoperative patients with severe underlying diseases (such as severe liver and kidney function, cardiopulmonary function, coagulation dysfunction, etc.)
  2. Patients with malignant tumors in other parts of the body

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ultra-low rectal cancer
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
the distance of intramural spread | 2023.01-2024.12

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Whenzhou Medical University, Wenzhou, Zhejiang, China